CLINICAL TRIAL: NCT03433755
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study to Evaluate Safety and Efficacy of Evolocumab (AMG 145) in Addition to Optimal Stable Background Statin Therapy in Chinese Subjects With Primary Hypercholesterolemia and Mixed Dyslipidemia
Brief Title: Safety and Efficacy of Evolocumab in Addition to Optimal Stable Background Statin Therapy in Chinese Participants With Primary Hypercholesterolemia and Mixed Dyslipidemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Prematurely Discontinued Amgen decision
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20150172
Record Dates: First submitted 2018-01-18; First posted 2018-02-15 (Actual); Results first posted 2021-08-20 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Primary Hypercholesterolemia; Mixed Dyslipidemia
Keywords: Evolocumab; Repatha; Statin; Chinese; China; Hypercholesterolemia; Mixed Dyslipidemia; High Cholesterol; Lowering cholesterol
MeSH Terms: conditions — Hypercholesterolemia | interventions — evolocumab

STUDY DESIGN:
Intervention Model Description: Participants will be screened for this study and if found eligible as described by the study protocol may be randomized into 1 of 4 groups. Randomized means that you are put into a group by chance. It is like drawing numbers out of a hat. Randomization will be done using a 2:2:1:1 ratio. This means for every 6 participants randomized:
  * 2 participants will be randomized to evolocumab 140 mg every 2 weeks
  * 2 participants will be randomized to evolocumab 420 mg once a month
  * 1 participant will be randomized to placebo every 2 weeks
  * 1 participant will be randomized to placebo once a month.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The dose frequencies of Q2W and QM will not be blinded but the identity of investigational product (evolocumab or matching SC placebo) will be blinded. In order to protect the blinding of the double-blind treatment period the following labs will be blinded post-investigational product treatment until unblinding of the clinical database and not reported to sites as noted below:
  • Blinded to the Amgen study team and site staff: lipid panel, Apolipoprotein A1 (ApoA1), Apolipoprotein B (ApoB), lipoprotein(a), high-sensitivity C-reactive protein (hs-CRP), and Proprotein convertase subtilisin/kexin type 9 (PCSK9).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Placebo Q2W (Placebo Comparator): Placebo subcutaneous (SC) Q2W for 12 weeks
  Interventions: Drug: placebo
- Placebo QM (Placebo Comparator): Placebo SC QM for 12 weeks
  Interventions: Drug: placebo
- Evolocumab 140 mg Q2W (Experimental): Evolocumab 140 mg SC Q2W for 12 weeks
  Interventions: Drug: evolocumab
- Evolocumab 420 mg QM (Experimental): Evolocumab 420 mg SC QM for 12 weeks
  Interventions: Drug: evolocumab

INTERVENTIONS:
Drug: evolocumab — Evolocumab will be administered per pre-filled auto-injector pen (AI/Pen). Participants will receive evolocumab (AMG 145) every 2 weeks or monthly subcutaneously.
  Other Names: Repatha; AMG 145
  Arms: Evolocumab 140 mg Q2W; Evolocumab 420 mg QM
Drug: placebo — Placebo will be administered per pre-filled auto-injector pen (AI/Pen). Participants will receive placebo every 2 weeks or monthly subcutaneously.
  Arms: Placebo Q2W; Placebo QM

SUMMARY:
This study is being done to learn more about evolocumab in Chinese people with primary hypercholesterolemia or mixed dyslipidemia. This study will see if evolocumab will reduce low density lipoprotein cholesterol (LDL-C) in Chinese people who are also taking a certain type of lipid-lowering medication (statins with or without ezetimibe) and whether it causes any side effects.

DETAILED DESCRIPTION:
This is a phase 3, multicenter, double-blind, randomized, placebo-controlled study of evolocumab in Chinese participants with hypercholesterolemia and mixed dyslipidemia. Participants who have signed the informed consent form (ICF) will have fasting lipids measured and all inclusion and exclusion criteria assessed. All eligible participants must be taking a maximum appropriate dose of an approved statin, not requiring up titration. Participants should maintain their current diet and exercise regimen.

Treatment and follow-up period will be 12 weeks with an additional phone call or other participant contact at week 14 for those receiving investigational product every 2 weeks (Q2W). The end of study (EOS) for participants on once monthly (QM) investigational product is at the week 12 visit, which must be at least 30 days post last dose of investigational product.

Evolocumab or placebo will be administered by self-injection under the skin at the study site or in an appropriate non-clinic setting (e.g., at home) by spring based prefilled auto injector/pen (AI/Pen). Participants must tolerate an injection of placebo with a prefilled auto injector/pen device to be used during the study prior to randomization.

Participants will be randomly added to 1 of 4 groups using a 2:2:1:1 ratio:

evolocumab 140 mg Q2W (86 participants total) evolocumab 420 mg QM (86 participants total) placebo Q2W (44 participants total) placebo QM (43 participants total). The dose frequencies of Q2W and QM will not be blinded but the identity of investigational product evolocumab or placebo will be blinded.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age at signing of informed consent form
* On an approved statin, with or without ezetimibe, at optimal stable daily dose(s) for at least 4 weeks before LDL-C screening and, in the opinion of the investigator, not requiring uptitration
* Fasting LDL-C as determined by central laboratory at screening ≥ 80 mg/dL
* Subject meets at least 1 of the following criteria for high/very high cardiovascular (CV) risk：

  * history of coronary artery disease
  * history of ischemic stroke
  * diagnosis of peripheral artery disease
  * an estimated glomerular filtration rate (eGFR) as determined by central laboratory at screening of ≥ 30 but < 60 ml/min/1.73m^2
  * diagnosis of diabetes mellitus type 2
  * presence of ≥ 3 of the following risk factors: ≥ 45 years of age if male; ≥ 55 years of age if female; hypertension; smoking; family history of premature cardiovascular disease (CVD; 1st degree of relative: male < 55 yr, female < 65 yr); high-density lipoprotein (HDL) cholesterol < 40 mg/dL; obesity (body mass index ≥ 28 kg/m^2)

OR

Subject does not meet high/very high CV risk criteria but fasting LDL-C as determined by central laboratory at screening ≥ 130 mg/dl

* Fasting triglycerides ≤ 400 mg/dL (4.5 mmol/L) by determined by central laboratory at screening
* Subject tolerates a screening placebo injection.

Exclusion Criteria:

* Myocardial infarction, unstable angina, percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG) or stroke within 3 months prior to randomization
* Planned coronary or other revascularization within 20 weeks of screening
* New York Heart Association (NYHA) III or IV heart failure, or last known left ventricular ejection fraction < 30
* Uncontrolled serious cardiac arrhythmia defined as recurrent and highly symptomatic ventricular tachycardia, atrial fibrillation with rapid ventricular response, or supraventricular tachycardia that are not controlled by medications, in the past 3 months prior to randomization
* Type 1 diabetes, new-onset (hemoglobin [Hb]A1c ≥ 6.5% or fasting plasma glucose (FPG) ≥ 126 mg/dL at screening without known diagnosis) or poorly controlled (HbA1c ≥ 8.5%) type 2 diabetes, as determined by central laboratory at screening
* Uncontrolled hypertension defined as sitting systolic blood pressure (SBP) > 180 mmHg or diastolic blood pressure (DBP) > 110 mmHg
* Subject has taken a cholesterylester transfer protein (CETP) inhibitor in the 12 months prior to randomization
* Subject has taken in the 6 weeks prior to LDL-C screening: red yeast rice, > 200 mg/day niacin, > 1000 mg/day omega-3 fatty acids (eg, dihydroxyacetone docosahexaenoic acid and eicosapentaenoic acid), stanols or prescription lipid-regulating drugs (eg, bile-acid sequestering resins, fibrates and derivatives) or other cholesterol lowering drugs or lipid-lowering dietary supplements or food additives other than statins and ezetimibe
* Treatment 3 months prior to LDL-C screening with any of the following drugs: systemic cyclosporine, systemic steroids, (intravenous [IV], intramuscular [IM], or by-mouth [PO]) (Note: hormone replacement therapy is permitted), vitamin A derivatives and retinol derivatives for the treatment of dermatologic conditions (eg, Accutane) (Note: vitamin A in a multivitamin preparation is permitted)
* Uncontrolled hypothyroidism or hyperthyroidism as defined by thyroid stimulating hormone (TSH) < 1.0 time the lower limit of normal (LLN) or > 1.5 times the upper limit of normal (ULN), respectively, at screening
* Severe renal dysfunction, defined as an eGFR < 30 ml/min/1.73m^2 at screening as estimated by Cockcroft-Gault method
* Active liver disease or hepatic dysfunction, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 times the ULN as determined by central laboratory analysis at screening
* Creatinine kinase (CK) > 5 times the ULN at screening
* Malignancy (except non-melanoma skin cancers, cervical in-situ carcinoma, breast ductal carcinoma in situ, or stage 1 prostate carcinoma) within the last 5 years prior to randomization
* Subject has previously received evolocumab or any other therapy to inhibit PCSK9
* Subject has known sensitivity to any of the active substances or their excipients to be administered during dosing, eg, carboxymethylcellulose
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the subject and investigator's knowledge.
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
* Currently receiving treatment in another investigational device or drug study, or less than 30 days before randomization since ending treatment on another investigational device or drug study(s) or planning to receive other investigational procedures while participating in this study
* Female subject of childbearing potential not willing to use an acceptable method(s) of effective birth control during treatment with investigational product and for an additional 15 weeks after the end of treatment with investigational product. Female subjects of non-childbearing potential who are not required to use contraception during the study and include those who have had a:

  * hysterectomy
  * bilateral salpingectomy
  * bilateral oophorectomy or
  * who are postmenopausal i. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. [A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy (HRT). However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

ii. Females on HRT and whose menopausal status is in doubt will be required to use one of the non-hormonal highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status before study enrollment.

Acceptable methods of effective birth control include:

* sexual abstinence (defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments; the reliability of sexual abstinence must be evaluated in relation to the duration of the trial and the preferred and usual lifestyle of the subject. [Periodic abstinence (eg., calendar, ovulation, symptothermal, postovulation methods), declaration of abstinence for the duration of a study, and withdrawal are not acceptable methods of contraception])
* bilateral tubal ligation/occlusion
* vasectomized partner (provided that partner is the sole sexual partner of the female subject of childbearing potential and that the vasectomized partner has received medical assessment of the surgical success)
* use of hormonal birth control methods (oral, intravaginal (eg. vaginal ring(s), transdermal, injectable, or implantable)
* intrauterine devices (IUDs)
* intrauterine hormonal releasing system (IUS)
* 2 barrier methods (each partner must use 1 barrier method) the male uses a condom and the female must choose either a diaphragm, OR cervical cap, OR contraceptive sponge with spermicide. If spermicide is not commercially available in the country or region, the 2 barrier method without spermicide is acceptable. (A female condom is not an option due to the risk of tearing when both partners use a condom.)

  * Female subject is pregnant or breast feeding (nursing), planning to become pregnant or planning to breastfeed (nurse) during treatment with investigational product and/or within 15 weeks after the end of treatment with investigational product.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (31):
- China (31):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou First PeoplesÂ Â Hospital, Guangzhou, Guangdong
  - Guangzhou Red Cross Hospital, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The Second Nanning Peoples Hospital, Nanning, Guangxi
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Wuhan Puai Hospital, Wuhan, Hubei
  - Changsha Central Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Inner Mongolia Peoples Hospital, Hohhot, Inner Mongolia
  - Suzhou Kowloon Hospital, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The Second Affiliated Hospital to Nanchang University, Nanchang, Jiangxi
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The Peoples Hospital of Liaoning Province, Shenyang, Liaoning
  - Jinan Central Hospital, Jinan, Shandong
  - Shanghai Yangpu District Central Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi An Jiao Tong University, Xi’an, Shanxi
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Fourth Centre Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Linhai, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Huashan Hospital Affiliated to Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Tan H, Li W, Huang Z, Han Y, Huang X, Li D, Xing X, Monsalvo ML, Wu Y, Mao J, Xin L, Chen J; HUA TUO study investigators. Efficacy and Safety of Evolocumab in Chinese Patients with Primary Hypercholesterolemia and Mixed Dyslipidemia: 12-Week Primary Results of the HUA TUO Randomized Clinical Trial. Cardiol Ther. 2023 Jun;12(2):341-359. doi: 10.1007/s40119-023-00304-x. Epub 2023 Feb 21. PMID 36802321
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 31 research centers in China from 09 May 2019 to 20 January 2020.
Pre-assignment Details: Participants were randomized 2:2:1:1 into the following treatment arms: evolocumab140 mg subcutaneously (SC) every 2 weeks (Q2W); evolocumab 420 mg SC once monthly (QM); placebo SC Q2W, or placebo SC QM. Randomization was stratified by entry cardiovascular (CV) risk (high/very high vs. not high/very high). Due to Human Genetic Resource Administration office of China (HGRAC) regulations/restrictions, 17 participants were not included in any analysis.
Period: Overall Study
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab 140 mg Q2W | Evolocumab 420 mg QM
Started | 42 | 41 | 79 | 80
Randomized and Treated | 41 | 41 | 79 | 80
Completed | 40 | 41 | 79 | 80
Not Completed | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Decision by Sponsor | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: All participants who were randomized and received at least 1 dose of study drug.
Groups:
- Placebo Q2W: Placebo SC Q2W for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab 140 mg Q2W | Evolocumab 420 mg QM | Total
Number analyzed (Participants) | 41 | 41 | 79 | 80 | 241
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (9.8) | 59.4 (10.9) | 61.2 (10.6) | 60.9 (9.8) | 60.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 28 | 29 | 78
  Male | 30 | 31 | 51 | 51 | 163
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 41 | 41 | 79 | 80 | 241
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 41 | 41 | 79 | 80 | 241
Stratification Factor: Cardiovascular (CV) Risk [Count of Participants; unit: Participants] — See eligibility criteria for the definition of high/very high cardiovascular (CV) risk. Participants not meeting high/very high CV risk criteria had fasting LDL-C as determined by central laboratory at screening ≥ 130 mg/dl.
  Participants
    High/Very High CV Risk | 37 | 38 | 73 | 74 | 222
    Not High/Very High CV Risk | 4 | 3 | 6 | 6 | 19
Low-Density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] | 120.9 (42.2) | 117.1 (28.2) | 113.7 (37.7) | 115.5 (30.1) | 116.1 (34.6)

OUTCOME MEASURES:

1. Primary Outcome: Co-Primary Endpoint: Percent Change From Baseline in LDL-C: Mean of Weeks 10 and 12
Description: Least squares mean is from the repeated measures linear effects model which includes treatment group, stratification factors, scheduled visit and the interaction of treatment with scheduled visit as covariates.
Time Frame: Baseline, Weeks 10 and 12
Population: Full Analysis Set: participants who were randomized and received at least 1 dose of study drug. Participants with baseline and post-baseline assessments.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Evolocumab 140 mg Q2W | Placebo QM | Evolocumab 420 mg QM
Number analyzed (Participants) | 37 | 69 | 35 | 71
percent change | 1.88 (3.72) | -68.86 (3.27) | -0.36 (3.78) | -70.10 (3.21)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Includes treatment group, stratification factors, scheduled visit and the interaction of treatment with scheduled visit as covariates; Treatment difference = -70.73, 95% CI 2-sided [-77.98 to -63.48], Standard Error of Mean 3.65 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab 420 mg QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -69.74, 95% CI 2-sided [-76.51 to -62.97], Standard Error of Mean 3.41 — Treatment difference = Evolocumab QM - Placebo QM

2. Primary Outcome: Co-Primary Endpoint: Percent Change From Baseline in LDL-C at Week 12
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Evolocumab 140 mg Q2W | Placebo QM | Evolocumab 420 mg QM
Number analyzed (Participants) | 34 | 64 | 27 | 66
percent change | 2.48 (4.18) | -68.39 (3.55) | 2.72 (4.25) | -63.09 (3.42)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -70.87, 95% CI 2-sided [-79.47 to -62.27], Standard Error of Mean 4.33 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab 420 mg QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -65.81, 95% CI 2-sided [-73.97 to -57.66], Standard Error of Mean 4.11 — Treatment difference = Evolocumab QM - Placebo QM

3. Secondary Outcome: Change From Baseline in LDL-C: Mean of Weeks 10 and 12
Description: as for outcome 1
Time Frame: Baseline, Weeks 10 and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo Q2W | Evolocumab 140 mg Q2W | Placebo QM | Evolocumab 420 mg QM
Number analyzed (Participants) | 37 | 69 | 35 | 71
mg/dL | -0.6 (5.4) | -77.1 (4.8) | -5.8 (5.8) | -83.0 (5.0)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -76.5, 95% CI 2-sided [-86.6 to -66.4], Standard Error of Mean 5.1 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab 420 mg QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -77.2, 95% CI 2-sided [-87.7 to -66.7], Standard Error of Mean 5.3 — Treatment difference = Evolocumab QM - Placebo QM

4. Secondary Outcome: Change From Baseline in LDL-C at Week 12
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo Q2W | Evolocumab 140 mg Q2W | Placebo QM | Evolocumab 420 mg QM
Number analyzed (Participants) | 34 | 64 | 27 | 66
mg/dL | -0.8 (5.8) | -76.7 (5.1) | -2.1 (6.1) | -75.1 (5.0)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -75.9, 95% CI 2-sided [-87.1 to -64.7], Standard Error of Mean 5.6 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab 420 mg QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -73.0, 95% CI 2-sided [-84.1 to -61.8], Standard Error of Mean 5.6 — Treatment difference = Evolocumab QM - Placebo QM

5. Secondary Outcome: Percent Change From Baseline in Non-High-Density Lipoprotein Cholesterol (Non-HDL-C): Mean of Weeks 10 and 12
Description: as for outcome 1
Time Frame: Baseline, Weeks 10 and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Evolocumab 140 mg Q2W | Placebo QM | Evolocumab 420 mg QM
Number analyzed (Participants) | 37 | 69 | 35 | 71
percent change | 2.36 (3.52) | -58.84 (3.10) | -0.06 (3.30) | -62.20 (2.81)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -61.20, 95% CI 2-sided [-68.04 to -54.37], Standard Error of Mean 3.44 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab 420 mg QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -62.15, 95% CI 2-sided [-67.97 to -56.32], Standard Error of Mean 2.94 — Treatment difference = Evolocumab QM - Placebo QM

6. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Evolocumab 140 mg Q2W | Placebo QM | Evolocumab 420 mg QM
Number analyzed (Participants) | 34 | 64 | 27 | 66
percent change | 3.86 (3.85) | -57.59 (3.30) | 1.78 (3.70) | -54.86 (2.99)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -61.45, 95% CI 2-sided [-69.25 to -53.65], Standard Error of Mean 3.93 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab 420 mg QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -56.65, 95% CI 2-sided [-63.66 to -49.63], Standard Error of Mean 3.54 — Treatment difference = Evolocumab QM - Placebo QM

7. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (ApoB): Mean of Weeks 10 and 12
Description: as for outcome 1
Time Frame: Baseline, Weeks 10 and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Evolocumab 140 mg Q2W | Placebo QM | Evolocumab 420 mg QM
Number analyzed (Participants) | 37 | 69 | 35 | 71
percent change | 1.80 (3.17) | -54.45 (2.79) | 0.07 (3.00) | -56.93 (2.54)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment Difference = -56.26, 95% CI 2-sided [-62.44 to -50.07], Standard Error of Mean 3.12 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab 420 mg QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment Difference = -57.00, 95% CI 2-sided [-62.35 to -51.65], Standard Error of Mean 2.70 — Treatment difference = Evolocumab QM - Placebo QM

8. Secondary Outcome: Percent Change From Baseline in ApoB at Week 12
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Evolocumab 140 mg Q2W | Placebo QM | Evolocumab 420 mg QM
Number analyzed (Participants) | 34 | 64 | 27 | 66
percent change | 2.53 (3.55) | -53.16 (3.03) | 1.20 (3.51) | -50.01 (2.77)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -55.69, 95% CI 2-sided [-62.98 to -48.41], Standard Error of Mean 3.67 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab 420 mg QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -51.21, 95% CI 2-sided [-58.06 to -44.37], Standard Error of Mean 3.45 — Treatment difference = Evolocumab QM - Placebo QM

9. Secondary Outcome: Percent Change From Baseline in Total Cholesterol: Mean of Weeks 10 and 12
Description: as for outcome 1
Time Frame: Baseline, Weeks 10 and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Evolocumab 140 mg Q2W | Placebo QM | Evolocumab 420 mg QM
Number analyzed (Participants) | 37 | 69 | 35 | 71
percent change | 1.32 (2.74) | -41.42 (2.42) | -0.09 (2.68) | -44.39 (2.28)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -42.74, 95% CI 2-sided [-48.06 to -37.41], Standard Error of Mean 2.68 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab 420 mg QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -44.30, 95% CI 2-sided [-49.02 to -39.58], Standard Error of Mean 2.38 — Treatment difference = Evolocumab QM - Placebo QM

10. Secondary Outcome: Percent Change From Baseline in Total Cholesterol at Week 12
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Placebo 420 mg SC QM: Placebo 420 mg SC QM for 12 weeks
Arm/Group | Placebo Q2W | Placebo 420 mg SC QM | Evolocumab 140 mg Q2W | Evolocumab 420 mg QM
Number analyzed (Participants) | 34 | 64 | 27 | 66
percent change | 2.69 (2.99) | -40.36 (2.57) | 1.17 (2.96) | -39.25 (2.40)
Statistical Analysis 1: Comparison: Placebo Q2W vs Placebo 420 mg SC QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -43.05, 95% CI 2-sided [-49.09 to -37.00], Standard Error of Mean 3.05 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Evolocumab 140 mg Q2W vs Evolocumab 420 mg QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -40.42, 95% CI 2-sided [-45.98 to -34.87], Standard Error of Mean 2.80 — Treatment difference = Evolocumab QM - Placebo QM

11. Secondary Outcome: Percentage of Participants With Target LDL-C < 70 mg/dL (1.8 mmol/L): Mean of Weeks 10 and 12
Description: Percentage of participants who were below the target LDL-C of 70 mg/dL (1.8 mmol/L) based on the mean LDL-C data collected at weeks 10 and 12.
Time Frame: Weeks 10 and 12
Population: Full Analysis Set: participants who were randomized and received at least 1 dose of study drug. Participants with observed data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Q2W | Evolocumab 140 mg Q2W | Placebo QM | Evolocumab 420 mg QM
Number analyzed (Participants) | 37 | 69 | 35 | 71
percentage of participants | 2.7 [0.5 to 13.8] | 89.9 [80.5 to 95.0] | 5.7 [1.6 to 18.6] | 97.2 [90.3 to 99.2]
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Based on Cochran Mantel Haenszel (CMH) test adjusted by the stratification factor; Treatment difference = 87.2, 95% CI 2-sided [72.6 to 92.8] — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab 420 mg QM; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Based on CMH test adjusted by the stratification factor; Treatment difference = 91.5, 95% CI 2-sided [76.9 to 96.1] — Treatment difference = Evolocumab QM - Placebo QM

12. Secondary Outcome: Percentage of Participants With Target LDL-C < 70 mg/dL (1.8 mmol/L) at Week 12
Time Frame: Week 12
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Q2W | Evolocumab 140 mg Q2W | Placebo QM | Evolocumab 420 mg QM
Number analyzed (Participants) | 34 | 64 | 27 | 66
percentage of participants | 0.0 [0.0 to 10.2] | 90.6 [81.0 to 95.6] | 3.7 [0.7 to 18.3] | 89.4 [79.7 to 94.8]
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Based on CMH test adjusted by the stratification factor; Treatment difference = 90.6, 95% CI 2-sided [76.6 to 95.6] — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab 420 mg QM; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Based on CMH test adjusted by the stratification factor; Treatment difference = 85.7, 95% CI 2-sided [68.2 to 91.9] — Treatment difference = Evolocumab QM - Placebo QM

13. Secondary Outcome: Percentage of Participants With LDL-C Response: Mean of Weeks 10 and 12
Description: Percentage of participants who had LDL-C response (50% reduction of LDL-C from baseline) based on the mean LDL-C using the data collected at weeks 10 and 12.
Time Frame: Baseline, Weeks 10 and 12
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Q2W | Evolocumab 140 mg Q2W | Placebo QM | Evolocumab 420 mg QM
Number analyzed (Participants) | 37 | 69 | 35 | 71
percentage of participants | 0.0 [0.0 to 9.4] | 87.0 [77.0 to 93.0] | 5.7 [1.6 to 18.6] | 94.4 [86.4 to 97.8]
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Based on CMH test adjusted by the stratification factor; Treatment difference = 87.0, 95% CI 2-sided [73.3 to 93.0] — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab 420 mg QM; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Based on CMH test adjusted by the stratification factor; Treatment difference = 88.7, 95% CI 2-sided [73.5 to 94.0] — Treatment difference = Evolocumab QM - Placebo QM

14. Secondary Outcome: Percentage of Participants With LDL-C Response (50% Reduction of LDL-C From Baseline) at Week 12
Description: LDL-C Response is defined as a 50% reduction of LDL-C from Baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Q2W | Evolocumab 140 mg Q2W | Placebo QM | Evolocumab 420 mg QM
Number analyzed (Participants) | 34 | 64 | 27 | 66
percentage of participants | 0.0 [0.0 to 10.2] | 82.8 [71.8 to 90.1] | 3.7 [0.7 to 18.3] | 86.4 [76.1 to 92.7]
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Based on CMH test adjusted by the stratification factor; Treatment difference = 82.8, 95% CI 2-sided [67.8 to 90.1] — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab 420 mg QM; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Based on CMH test adjusted by the stratification factor; Treatment difference = 82.7, 95% CI 2-sided [64.8 to 89.7] — Treatment difference = Evolocumab QM - Placebo QM

15. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) [Lp(a)]: Mean of Weeks 10 and 12
Description: as for outcome 1
Time Frame: Baseline, Weeks 10 and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Evolocumab 140 mg Q2W | Placebo QM | Evolocumab 420 mg QM
Number analyzed (Participants) | 37 | 69 | 35 | 71
percent change | 4.96 (4.97) | -43.49 (4.46) | 11.27 (4.37) | -29.16 (3.58)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -48.45, 95% CI 2-sided [-57.78 to -39.11], Standard Error of Mean 4.71 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab 420 mg QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -40.43, 95% CI 2-sided [-48.62 to -32.24], Standard Error of Mean 4.13 — Treatment difference = Evolocumab QM - Placebo QM

16. Secondary Outcome: Percent Change From Baseline in Lp(a) at Week 12
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Evolocumab 140 mg Q2W | Placebo QM | Evolocumab 420 mg QM
Number analyzed (Participants) | 34 | 64 | 27 | 66
percent change | 1.87 (5.21) | -42.83 (4.60) | 14.53 (5.64) | -23.73 (4.18)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -44.70, 95% CI 2-sided [-54.76 to -34.65], Standard Error of Mean 5.07 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab 420 mg QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -38.26, 95% CI 2-sided [-49.94 to -26.59], Standard Error of Mean 5.88 — Treatment difference = Evolocumab QM - Placebo QM

17. Secondary Outcome: Percent Change From Baseline in Triglycerides: Mean of Weeks 10 and 12
Description: as for outcome 1
Time Frame: Baseline, Weeks 10 and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Evolocumab 140 mg Q2W | Placebo QM | Evolocumab 420 mg QM
Number analyzed (Participants) | 37 | 69 | 35 | 71
percent change | 5.23 (4.77) | -9.86 (4.19) | 3.03 (4.85) | -16.64 (4.09)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority; p = 0.008, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -15.09, 95% CI 2-sided [-24.44 to -5.75], Standard Error of Mean 4.71 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab 420 mg QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -19.67, 95% CI 2-sided [-28.30 to -11.05], Standard Error of Mean 4.35 — Treatment difference = Evolocumab QM - Placebo QM

18. Secondary Outcome: Percent Change From Baseline in Triglycerides at Week 12
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Evolocumab 140 mg Q2W | Placebo QM | Evolocumab 420 mg QM
Number analyzed (Participants) | 34 | 64 | 27 | 66
percent change | 10.01 (5.63) | -7.55 (4.73) | 0.69 (5.56) | -11.66 (4.37)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority; p = 0.008, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -17.56, 95% CI 2-sided [-29.42 to -5.69], Standard Error of Mean 5.98 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab 420 mg QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -12.35, 95% CI 2-sided [-23.04 to -1.67], Standard Error of Mean 5.38 — Treatment difference = Evolocumab QM - Placebo QM

19. Secondary Outcome: Percent Change From Baseline in High-Density Lipoprotein Cholesterol (HDL-C): Mean of Weeks 10 and 12
Description: as for outcome 1
Time Frame: Baseline, Weeks 10 and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Evolocumab 140 mg Q2W | Placebo QM | Evolocumab 420 mg QM
Number analyzed (Participants) | 37 | 69 | 35 | 71
percent change | 1.01 (2.65) | 9.45 (2.35) | 1.86 (2.60) | 8.66 (2.18)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority; p = 0.008, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = 8.44, 95% CI 2-sided [3.35 to 13.52], Standard Error of Mean 2.56 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab 420 mg QM; Test type: Superiority; p = 0.017, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = 6.80, 95% CI 2-sided [2.10 to 11.50], Standard Error of Mean 2.37 — Treatment difference = Evolocumab QM - Placebo QM

20. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 12
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Evolocumab 140 mg Q2W | Placebo QM | Evolocumab 420 mg QM
Number analyzed (Participants) | 34 | 64 | 27 | 66
percent change | 1.95 (2.88) | 9.89 (2.49) | 0.95 (2.97) | 7.12 (2.33)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority; p = 0.008, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = 7.94, 95% CI 2-sided [2.18 to 13.71], Standard Error of Mean 2.91 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab 420 mg QM; Test type: Superiority; p = 0.017, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = 6.17, 95% CI 2-sided [0.42 to 11.92], Standard Error of Mean 0.036 — Treatment difference = Evolocumab QM - Placebo QM

21. Secondary Outcome: Percent Change From Baseline in Very Low-Density Lipoprotein Cholesterol (VLDL-C): Mean of Weeks 10 and 12
Description: as for outcome 1
Time Frame: Baseline, Weeks 10 and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Evolocumab 140 mg Q2W | Placebo QM | Evolocumab 420 mg QM
Number analyzed (Participants) | 37 | 69 | 35 | 71
percent change | 7.08 (5.32) | -15.88 (4.73) | 4.95 (4.97) | -22.87 (4.21)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority; p = 0.0002, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -22.96, 95% CI 2-sided [-33.12 to -12.81], Standard Error of Mean 4.44 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab 420 mg QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -27.81, 95% CI 2-sided [-36.60 to -19.02], Standard Error of Mean 4.44 — Treatment difference = Evolocumab QM - Placebo QM

22. Secondary Outcome: Percent Change From Baseline in VLDL-C at Week 12
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Evolocumab 140 mg Q2W | Placebo QM | Evolocumab 420 mg QM
Number analyzed (Participants) | 34 | 64 | 27 | 66
percent change | 11.23 (6.12) | -10.55 (5.22) | 1.72 (5.57) | -14.02 (4.42)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority; p = 0.0002, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -21.78, 95% CI 2-sided [-34.31 to -9.25], Standard Error of Mean 6.32 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab 420 mg QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; Treatment difference = -15.74, 95% CI 2-sided [-26.31 to -5.18], Standard Error of Mean 5.33 — Treatment difference = Evolocumab QM - Placebo QM

ADVERSE EVENTS:
Time Frame: Mortality: from randomization to end of study (EOS) date; median (min, max) duration was 3.22 (0.99, 4.01) months. AEs: from first dose up to last dose + 30 days or EOS date, whichever was earlier; median (min, max) duration was 2.86 (1.02, 3.88) months.
Description: Mortality is reported for randomized participants. Serious and other AEs are reported for randomized participants who received at least one dose of study drug.
Groups:
- Placebo QM: Placebo SC Q2W for 12 weeks
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab 140 mg Q2W | Evolocumab 420 mg QM
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/41 | 0/79 | 0/80
Serious Adverse Events (participants affected / at risk) | 2/41 | 4/41 | 6/79 | 1/80
Other Adverse Events (participants affected / at risk) | 22/41 | 22/41 | 45/79 | 42/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=41) | Placebo QM (N=41) | Evolocumab 140 mg Q2W (N=79) | Evolocumab 420 mg QM (N=80)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1 | 0
Goitre (Endocrine disorders) | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=41) | Placebo QM (N=41) | Evolocumab 140 mg Q2W (N=79) | Evolocumab 420 mg QM (N=80)
Abnormal clotting factor (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiomegaly (Cardiac disorders) | 0 | 0 | 1 | 0
Left atrial enlargement (Cardiac disorders) | 0 | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 2 | 0 | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0
Goitre (Endocrine disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Chest discomfort (General disorders) | 0 | 0 | 1 | 0
Facial pain (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Feeling cold (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 3 | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Congestive hepatopathy (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Gallbladder polyp (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic mass (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 2 | 3 | 1
Liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Helicobacter infection (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 1
Syphilis (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 2 | 7 | 6
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 2
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 0
Bacterial test (Investigations) | 0 | 0 | 1 | 0
Bacterial test positive (Investigations) | 0 | 0 | 1 | 0
Bilirubin conjugated increased (Investigations) | 1 | 0 | 0 | 0
Blood alkaline phosphatase (Investigations) | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 1 | 1
Blood bilirubin unconjugated increased (Investigations) | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 1
Blood pressure increased (Investigations) | 0 | 0 | 3 | 0
Blood urea increased (Investigations) | 1 | 0 | 1 | 1
Body temperature increased (Investigations) | 0 | 0 | 1 | 0
Carotid intima-media thickness increased (Investigations) | 0 | 1 | 0 | 0
Glucose urine present (Investigations) | 1 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0
Protein urine present (Investigations) | 0 | 0 | 4 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0
Urinary occult blood positive (Investigations) | 0 | 0 | 3 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 1
White blood cells urine positive (Investigations) | 0 | 0 | 3 | 0
pH urine increased (Investigations) | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypovitaminosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Carotid arteriosclerosis (Nervous system disorders) | 0 | 1 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 1 | 0
Microalbuminuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Renal cyst (Renal and urinary disorders) | 1 | 0 | 2 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Breast swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Prostatic calcification (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0
Blood pressure inadequately controlled (Vascular disorders) | 0 | 1 | 3 | 0
Hypertension (Vascular disorders) | 1 | 3 | 6 | 4
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0
Vascular wall hypertrophy (Vascular disorders) | 0 | 0 | 2 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2016-06-06): https://cdn.clinicaltrials.gov/large-docs/55/NCT03433755/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/55/NCT03433755/SAP_001.pdf